CLINICAL TRIAL: NCT07200440
Title: Comparative Accuracy of Conventional Scan Bodies, Intra-oral Photogrammetry, and Calibrated Scan Flags in Full-Arch Implant Scanning: An In-Vitro Study
Brief Title: Comparative Accuracy of Conventional Scan Bodies, Intra-oral Photogrammetry, and Calibrated Scan Flags in Full-Arch Implant Scanning
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed El Saharty, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Mohamed El Saharty Scan
Record Dates: First submitted 2025-02-20; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Accuracy of Different Scanning Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- conventional scan bodies (Active Comparator): Digital scans using conventional scan bodies scanned with a desktop scanner.
  Interventions: Procedure: Control
- scan bodies scanned with an intra-oral scanner (Experimental): Digital scans using conventional scan bodies scanned with an intra-oral scanner.
  Interventions: Procedure: Intervention 1
- intra-oral photogrammetry (Experimental): Digital scans using intra-oral photogrammetry scanned with an intra-oral scanner.
  Interventions: Procedure: Intervention 2
- calibrated scan flags (Experimental): Digital scans using calibrated scan flags scanned with an intra-oral scanner.
  Interventions: Procedure: Intervention 3

INTERVENTIONS:
Procedure: Intervention 1 — Digital scans using conventional scan bodies scanned with an intra-oral scanner.
  Arms: scan bodies scanned with an intra-oral scanner
Procedure: Intervention 2 — Digital scans using intra-oral photogrammetry scanned with an intra-oral scanner.
  Arms: intra-oral photogrammetry
Procedure: Intervention 3 — Digital scans using calibrated scan flags scanned with an intra-oral scanner.
  Arms: calibrated scan flags
Procedure: Control — Digital scans using conventional scan bodies scanned with a desktop scanner.
  Arms: conventional scan bodies

SUMMARY:
To assess and compare the accuracy of digital scans obtained using three different scanning protocols -conventional scan bodies, Intra-oral photogrammetry, and calibrated scan flags- on completely edentulous dental model with full-arch implants.

DETAILED DESCRIPTION:
Digital scans have revolutionized prosthetic workflows by offering increased efficiency and accuracy compared to conventional techniques . Studies highlight that their accuracy depends on the scanning protocol and equipment used. Conventional scan bodies, which are well-established and commonly used for digital scans, are generally reliable; however, their accuracy can be influenced by factors such as angulation, the number of implants, and the scanning technique. Intra-oral photogrammetry has gained attention for its ability to accurately record implant positions without relying on physical scan bodies . Many systems utilize this technology to improve accuracy, particularly in complex full-arch cases, though direct comparisons with other methods remain limited. Calibrated Scan Flags represent a novel approach, incorporating enhanced features to reduce errors associated with angulation and improve the capture of implant positions. While initial studies suggest improved precision, further comparative data are required . Previous research comparing these methods often focuses on isolated factors, such as time efficiency or user preferences, with limited emphasis on accuracy. Therefore, a direct comparative analysis of these three scanning protocols is needed to address this gap.

ELIGIBILITY:
Inclusion Criteria:

* Edentulous dental model simulating completely edentulous patients.
* Model containing full-arch implant analogs placed in standardized positions.
* Access to compatible scan bodies for all three scanning protocols.

Exclusion Criteria:

* Dental models with defects, such as fractures or irregularities, that may influence scanning accuracy.
* Implant analogs placed at non-standardized or inconsistent angles.
* Scan bodies or equipment showing signs of wear or damage that could compromise results.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Accuracy of multiunit abutment positions | 7 days
  positions and angles of the multiunit abutments

IPD SHARING:
Plan to Share IPD: Undecided
Will be decided after getting the results

REFERENCES:
- [Background] Ma B, Yue X, Sun Y, Peng L, Geng W. Accuracy of photogrammetry, intraoral scanning, and conventional impression techniques for complete-arch implant rehabilitation: an in vitro comparative study. BMC Oral Health. 2021 Dec 10;21(1):636. doi: 10.1186/s12903-021-02005-0. PMID 34893053
- [Background] Buzayan M, Baig MR, Yunus N. Evaluation of accuracy of complete-arch multiple-unit abutment-level dental implant impressions using different impression and splinting materials. Int J Oral Maxillofac Implants. 2013 Nov-Dec;28(6):1512-20. doi: 10.11607/jomi.2958. PMID 24278919